CLINICAL TRIAL: NCT05468853
Title: Manipulating the Reward Circuit With TMS
Brief Title: Reward Circuit Targeted iTBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Derek Nee, Associate Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00002776; R21MH129653 (NIH)
Record Dates: First submitted 2022-07-01; First posted 2022-07-21 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Transcranial Magnetic Stimulation
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- rmPFC-iTBS (Experimental): Transcranial magnetic stimulation delivered to the rostral medial prefrontal cortex. 600 pulses delivered in 50 Hz bursts every 5 Hz for 2 seconds followed by 8 seconds of no stimulation repeated 20 times at 80% of resting motor threshold. Repeated daily for 5 consecutive days.
  Interventions: Device: transcranial magnetic stimulation
- Inion-iTBS (Active Comparator): Transcranial magnetic stimulation delivered to the inion. 600 pulses delivered in 50 Hz bursts every 5 Hz for 2 seconds followed by 8 seconds of no stimulation repeated 20 times at 80% of resting motor threshold. Repeated daily for 5 consecutive days.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation delivered to the scalp targeting medial prefrontal cortex
  Arms: rmPFC-iTBS
Device: transcranial magnetic stimulation — Transcranial magnetic stimulation delivered to the inion
  Arms: Inion-iTBS

SUMMARY:
The objective of this study is to examine the effect of intermittent theta-burst transcranial magnetic stimulation (iTBS) targeting the reward circuit.

DETAILED DESCRIPTION:
The study will examine the effect of medial prefrontal cortex (MPFC)-iTBS on the reward circuit, reward sensitivity, and anhedonia. The reward circuit will be assessed using functional MRI (fMRI) connectivity and activation during the Doors Task. Reward sensitivity will be assessed using an event-related potential called the reward positivity or RewP. The RewP will be measured using electroencephalography (EEG) during the Doors Task. Anhedonia will be measured using the Dimensional Anhedonia Ratings Scale (DARS).

The Doors Task was designed to examine reward processing in a simple, well-controlled paradigm. On each trial, participants select one of two doors. Gain (50 cents) or loss (25 cents) feedback is provided. Gains elicit a positive potential referred to as the RewP, while losses elicit a negative potential referred to as the feedback reward negativity (FRN). Gains also show increased activation in reward-related brain areas (e.g. ventral striatum) relative to losses in the fMRI signal.

Each participant will complete a baseline session including structural MRI, fMRI and EEG during the Doors task, and transcranial magnetic stimulation (TMS) motor thresholding. The ventral striatum (VS) will be identified on the structural MRI. The MPFC will be identified as a rostral-medial cortical area in prefrontal cortex with high connectivity to the VS. A control site, inion, will be identified using visual inspection of the skull.

Each participant will complete 2 weeks of iTBS sessions. Each week will target a different site (experimental: MPFC; control: inion). iTBS will be performed once a day for 5 consecutive days at each site, with order counter-balanced across participants in a cross-over design. 1 week of washout will follow each week of iTBS. At the end of each week, participants will perform the Doors task while being measured with EEG, and complete the DARS. At the end of the iTBS weeks, participants will also perform the Doors task while being measured with fMRI.

fMRI activation of the MPFC target and VS, and VS-MPFC fMRI connectivity will be compared at baseline, following the MPFC-iTBS week, and following the control-iTBS week. Changes specific to MPFC-iTBS will provide evidence of the effect of MPFC-iTBS on the reward circuit. The RewP and DARS will be compared at baseline, and after each week, respectively. Changes specific to MPFC-iTBS will provide evidence of the effect of MPFC-iTBS on the reward sensitivity and anhedonia. Changes that persist following washout will provide an indication of a lasting effect of MPFC-iTBS.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Native English speaker or fluent by the age of 6
* Elevated self-reported anhedonia

Exclusion Criteria:

* Left-handed
* Metal in head
* Brain tumor, stroke, aneurysm, multiple sclerosis
* Active substance use disorder in last 3 months
* Dementia or other cognitive disorder making unable to engage in treatment
* History or diagnosis of schizophrenia, schizoaffective disorder, delusional disorder, or other psychiatic illness that precludes safe participation in trial
* Suicidal risk that precludes safe participation
* obsessive-compulsive disorder
* Inability to stop taking any mediation that significant lowers the seizure threshold (e.g. tricyclic antidepressants, clozapine, etc.)
* Severe traumatic brain injury
* Non-English speaker

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- FSU MRI Facility, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Behavioral and imaging data will be shared
Supporting Information: Analytic Code
Time Frame: Within a year following publication of findings
Access Criteria: Behavioral and imaging data will be accessible from https://nda.nih.gov/edit_collection.html?id=4341 by NDA users

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants complete 1) a baseline functional MRI scan to determine targets for transcranial magnetic stimulation (TMS), and 2) motor thresholding to determine intensity of TMS. Participants are not assigned to arms if they cannot perform the task inside the MRI scanner (e.g. due to claustrophobia), if they cannot tolerate TMS (e.g., due to discomfort), and if they have contraindications for MRI or TMS (e.g., pro-epileptic medications, neurological conditions).
Groups:
- rmPFC-iTBS Then Inion-iTBS: Transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance. Each visit consists of 600 pulses delivered in 2 second trains of 50 Hz bursts every 5 Hz with 8 seconds in-between trains at 80% of resting motor threshold to one target. For a given target, stimulation was performed once a day for 5 consecutive days. A 9 day washout period followed prior to stimulating the alternate target. This arm completed transcranial magnetic stimulation to the rostromedial prefrontal cortex (rmPFC) first followed by the inion.
- Inion-iTBS Then rmPFC-iTBS: Transcranial magnetic stimulation: Transcranial magnetic stimulation delivered to the scalp targeting specific brain structures via stereotactic guidance. Each visit consists of 600 pulses delivered in 2 second trains of 50 Hz bursts every 5 Hz with 8 seconds in-between trains at 80% of resting motor threshold to one target. For a given target, stimulation was performed once a day for 5 consecutive days. A 9 day washout period followed prior to stimulating the alternate target. This arm completed transcranial magnetic stimulation to the inion first followed by the rostromedial prefrontal cortex (rmPFC).
Period: Overall Study
Arm/Group | rmPFC-iTBS Then Inion-iTBS | Inion-iTBS Then rmPFC-iTBS
Started | 35 | 34
Completed | 28 | 28
Not Completed | 7 | 6
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — incidental MRI finding | 1 | 2
Not completed — could not tolerate rmPFC-iTBS | 3 | 2
Not completed — illness | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rmPFC-iTBS Then Inion-iTBS | Inion-iTBS Then rmPFC-iTBS | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.5143 (6.38183) | 24.1176 (9.22041) | 23.8116 (7.85582)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 26 | 48
  Male | 13 | 8 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 21 | 25 | 46
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 28 | 29 | 57
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Anhedonia Post-intervention and Washout
Description: change in self-reported anhedonia from baseline averaged across post-intervention and post-washout measured using the score on the Dimensional Anhedonia Rating Scale (DARS); score range is 0-68 with higher scores meaning better outcomes (less anhedonia)
Time Frame: baseline, one-hour post-intervention, one-week post-intervention
Population: 4 participants with incomplete data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 52 | 52
Scores on a scale | 6.4231 (1.4585) | 5.4327 (1.1042)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.0452, t-test, 1 sided; Adjusted for stimulation order

2. Primary Outcome: Change in Anhedonia Post-intervention
Description: change in self-reported anhedonia from baseline immediately following the intervention measured using the score on the Dimensional Anhedonia Rating Scale (DARS); score range is 0-68 with higher scores meaning better outcomes (less anhedonia)
Time Frame: baseline, 1 hour post-intervention
Population: 4 participants with incomplete data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 52 | 52
Scores on a scale | 5.8462 (1.4558) | 4.75 (1.1042)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.1182, t-test, 1 sided; Adjusted for stimulation order

3. Primary Outcome: Change in Anhedonia Post-washout
Description: change in self-reported anhedonia from baseline following a week of washout post-intervention measured using the score on the Dimensional Anhedonia Rating Scale (DARS); score range is 0-68 with higher scores meaning better outcomes (less anhedonia)
Time Frame: baseline, 1 week post-intervention
Population: 4 participants with incomplete data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 52 | 52
Scores on a scale | 7 (1.5696) | 6.1154 (1.3255)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.1861, t-test, 1 sided; Adjusted for stimulation order

4. Primary Outcome: Change in RewP Post-intervention and Washout Measured Via EEG
Description: change in reward positivity from baseline averaged across immediately post-intervention and post-washout assessed via the EEG event-related potential (ERP) to feedback over FCz in microvolts
Time Frame: baseline, immediately post-intervention, one-week post-intervention
Population: 3 participants who had incomplete data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 53 | 53
microvolts | 0.2027 (0.6153) | -0.3760 (0.6280)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.1380, t-test, 1 sided; Adjusted for stimulation order

5. Secondary Outcome: Change in Reward Activation Measured Via fMRI
Description: Change in reward-related activation in the ventral striatum assessed via the fMRI blood-oxygenation level dependent (BOLD) signal following feedback (arbitrary units). More positive values indicate greater activation relative to baseline (more reward-related signal).
Time Frame: baseline, 15 minutes post-intervention
Population: 8 participants who had excessive head motion (root-mean square of framewise displacement > 0.3) were not analyzed. 2 participants with missing data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: arbitrary units
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 46 | 46
arbitrary units | -0.1067 (0.1315) | -0.0702 (0.1024)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.71946, ANOVA; Adjusted for stimulation order

6. Secondary Outcome: Change in Reward Connectivity Measured Via fMRI
Description: Change in fMRI connectivity between ventral striatum and medial prefrontal cortex assessed via correlations in the fMRI blood-oxygenation level dependent (BOLD) signal between these areas (z-scored correlation coefficient). More positive values indicate more positive correlations in BOLD signals between the ventral striatum and medial prefrontal cortex relative to baseline.
Time Frame: baseline, 15 minutes post-intervention
Population: 10 participants who had excessive head motion (root-mean square of framewise displacement > 0.3 in any visit) were not analyzed. 2 participants with missing data were not analyzed. 16 participants who did not complete the study were not analyzed.
Measure: Mean (Standard Error); unit: z-scored correlation coefficient
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 44 | 44
z-scored correlation coefficient | -0.0463 (0.0275) | 0.0049 (0.0261)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.19941, ANOVA; Adjusted for stimulation order

7. Primary Outcome: Change in RewP Post-intervention Measured Via EEG
Description: change in reward positivity from baseline immediately following the intervention assessed via the EEG event-related potential (ERP) to feedback over FCz in microvolts
Time Frame: baseline, immediately post-intervention
Population: as for outcome 4
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 53 | 53
microvolts | 0.3579 (0.7129) | -0.2191 (0.7721)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.1969, t-test, 1 sided; Adjusted for stimulation order

8. Primary Outcome: Change in RewP Post-washout Measured Via EEG
Description: change in reward positivity from baseline immediately following a week of washout post-intervention assessed via the EEG event-related potential (ERP) to feedback over FCz in microvolts
Time Frame: baseline, 1 week post-intervention
Population: as for outcome 4
Measure: Mean (Standard Error); unit: microvolts
Arm/Group | rmPFC-iTBS | Inion-iTBS
Number analyzed (Participants) | 53 | 53
microvolts | 0.0475 (0.8218) | -0.5328 (0.7189)
Statistical Analysis 1: Comparison: rmPFC-iTBS vs Inion-iTBS; Test type: Superiority; p = 0.2536, t-test, 1 sided; Adjusted for stimulation order

ADVERSE EVENTS:
Time Frame: From enrollment until the end of washout, up to 5 weeks
Arm/Group | rmPFC-iTBS Then Inion-iTBS | Inion-iTBS Then rmPFC-iTBS
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
Due to a programming error, the rmPFC was mistargeted in 55 participants. For these participants, stimulation of the rmPFC was weaker than intended. This issue may have undermined the efficacy of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-07-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT05468853/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/53/NCT05468853/ICF_001.pdf